CLINICAL TRIAL: NCT04031807
Title: Risk Factors for Failure After Single-incision Sling Procedure. Retrospective Analysis of 132 Women
Brief Title: Risk Factors for Failure After Single-incision Sling Procedure in Women With Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Sponsor
Other Study IDs: MaltepeU1
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Stress Urinary Incontinence
Keywords: Single-Incision Sling; Stress Urinary Incontinence; Failure
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Single-Incision Sling — The women with stress urinary incontinence underwent single-incision sling procedure.

SUMMARY:
The main risk factors for failure after single-incision slings are reduced urethral mobility and stress urinary incontinence severity in long-term follow-up.

DETAILED DESCRIPTION:
The medical records of the 132 patients were retrospectively analyzed. Preoperative assessment included medical history and urogynecological examination. Patients were asked to answer validated questionnaires such as Urinary Distress Inventory (UDI-6) and Incontinence Impact Questionnaire (IIQ-7). Objective cure of SUI was defined as the absence of demonstrable leakage of urine on the cough stress test. Subjective cure was based on negative response to UDI-6, question 3. Patients were divided according to objective cure rate into two groups: cured (Group A) and failed patients (Group B).

ELIGIBILITY:
Inclusion Criteria:

Women who underwent single-incision sling procedure for stress urinary incontinence

Exclusion Criteria:

Urodinamically proven detrusor overactivity

Neurogenic bladder

Previous anti-incontinence surgery including midurethral slings

Postvoidal residual volume (PVR) >100mL

Previous radical pelvic surgery

Anterior pelvic organ prolapse greater than stage I

Ages: 37 Years to 78 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: From September 2009 to September 2017, the medical records of the patients who underwentsingle-incision sling procedure for stress urinary incontinence without concomitant pelvic prolapse surgery were analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
objective cure | September 2009 to September 2017
  negative cough stress test

SECONDARY OUTCOMES:
subjective cure | September 2009 to September 2017
  negative response to Urinary Distress Inventory (UDI-6), question 3.

CONTACTS AND LOCATIONS:
Overall Officials: BERNA HALILOGLU PEKER, PROFESSOR, Principal Investigator — MALTEPE UNIVERSITY FACULTY OF MEDICINE DEPARTMENT OF OB&GYN
Locations (1):
- Maltepe University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No